CLINICAL TRIAL: NCT06962644
Title: Association of Urinary Tract Infection With Preeclampsia During Pregnancy
Status: Recruiting | Type: Observational
Sponsor: Pakistan Air Force (PAF) Hospital Islamabad (Other)
Responsible Party: Principal Investigator, Wajeeha Fatima, Principal Investigator, Pakistan Air Force (PAF) Hospital Islamabad
Other Study IDs: TrialUTI
Record Dates: First submitted 2025-04-22; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Urinary Tract Infection (Diagnosis); Preeclampsia
Keywords: Preeclampsia; Pregnancy; Urinary tract infection; Term Birth
MeSH Terms: conditions — Urinary Tract Infections; Disease; Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- UTI exposed: Patients suffering from UTI as per protocol
  Interventions: Other: Preeclampsia developed
- UTI non exposed: Patients having no clinical and laboratory evidence of UTI
  Interventions: Other: Preeclampsia developed

INTERVENTIONS:
Other: Preeclampsia developed — Preecalmpsia will be defined as per study protocol
  Other Names: preeclampsia not developed

SUMMARY:
Urinary tract infections (UTIs) are a major clinical issue, especially in pregnant women, due to physiological changes that increase susceptibility. If untreated, UTIs can lead to severe complications like preterm labor and low birth weight. Preeclampsia, a hypertensive disorder affecting 0.2-9.2% of pregnancies, is another leading cause of maternal and fetal complications. The relationship between UTIs and preeclampsia remains controversial, with some studies suggesting an association while others show conflicting results. Research gaps highlight the need for region-specific studies, particularly in Pakistan, where both conditions contribute significantly to maternal and neonatal morbidity.

This study aims to investigate the association between UTIs and preeclampsia in pregnant women in Pakistan. It will use a cohort design, enrolling 160 patients (80 with UTIs, 80 without) from the Obstetrics Department of PAF Hospital, Islamabad. Participants will be followed until delivery, with preeclampsia diagnosed based on blood pressure and proteinuria criteria. Data will be analyzed using SPSS to calculate relative risk (RR), with statistical significance set at RR >1 and p ≤ 0.05. The findings could help improve prenatal care and reduce adverse outcomes in high-risk populations.

DETAILED DESCRIPTION:
INTRODUCTION Urinary tract infections (UTIs) are a significant clinical concern, representing one of the most common bacterial infections in women, particularly during pregnancy. Globally, UTIs account for a substantial proportion of healthcare visits and are implicated in severe complications, including maternal and neonatal morbidity. The physiological and anatomical changes that occur during pregnancy, such as urinary stasis, hormonal influences, and alterations in the immune system, increase susceptibility to both asymptomatic bacteriuria and symptomatic UTIs. These infections can escalate to severe outcomes if untreated, with potential risks to maternal and fetal health, including preterm labor, low birth weight, and perinatal mortality. Concurrently, preeclampsia, a hypertensive disorder of pregnancy, which 0.2 to 9.2% of pregnancies, remains a leading cause of maternal and fetal complications. With its multifactorial etiology involving placental ischemia, systemic inflammation, and endothelial dysfunction, preeclampsia poses a critical challenge in obstetric care.

The relationship between UTIs and preeclampsia is an area of considerable clinical interest yet remains controversial. While some studies have highlighted an association between maternal infections, including UTIs, and an increased risk of preeclampsia, others have yielded conflicting results. Factors such as immune system dysregulation, systemic inflammation, and endothelial dysfunction, which are central to preeclampsia, may be exacerbated by UTIs. Despite extensive research, inconsistencies in prevalence estimates, study designs, and patient populations have hindered a definitive understanding of this association. One study found that 40% and 17.5% patients developed preeclampsia with and without UTI exposure respectively (p value 0.036). The relative risk (RR) was 2.47 (95%CI 1.1789 to 5.1777) with p value of 0.0166. Another study showed that UTI increases the risk of preeclampsia the OR was significant, but RR was not significant. [OR=1.86, (95% Confidence: 2.235-1.608) (p<0.043), RR 1.2028 (95%CI 0.9018 to 1.6041, p = 0.2089).

The results of a study showed that among 393 pregnant women enrolled, 110 (28.0%), had significant bacteriuria and women with preeclampsia had 7.7 odds of having significant bacteriuria (p-value <0.001). Radu, V. D., et al. found that there was no association of UTI and preeclampsia (aOR 2.07 with 95% CI 0.63-6.65, P value = 0.22). These knowledge gaps underscore the need for region-specific studies to assess whether UTIs contribute to preeclampsia and how they might influence maternal and perinatal outcomes, particularly in populations with distinct socioeconomic, healthcare, and environmental factors.

This study aims to investigate the association between UTIs and preeclampsia during pregnancy in Pakistan, where both conditions significantly contribute to maternal and neonatal morbidity and mortality. Pakistan's high burden of maternal infections and hypertensive disorders of pregnancy necessitates targeted research to identify preventable risk factors and improve clinical outcomes. 3, 6 By exploring the interplay between UTIs and preeclampsia, this research seeks to provide evidence-based insights that can inform public health strategies, enhance prenatal care protocols, and ultimately reduce the adverse effects of these conditions on maternal and fetal health in this region.

OBJECTIVE To find association of urinary traction infection with preeclampsia in pregnancy.

OPERATIONAL DEFINITIONS Urinary tract infection (UTI): It will be defined as >15 pus cells/high power field (HPF) in clean catch midstream urine after centrifugation and sedimentation.

Preeclampsia: It will be defined as BP >140/90 mmHg on minimum two occasions after 20 weeks of pregnancy alongside presence of proteinuria (≥300 mg/day or at least 1+ dipstick testing or spot urine protein/creatinine ratio of ≥30 mg/mmol).

HYPOTHESIS There is an association of urinary traction infection with preeclampsia in pregnancy.

METHODS AND MATERIALS Study design: Cohort study. Setting: Obstetrics and Gynecology Department, PAF Hospital, Islamabad. Duration of study: The study will be completed in a minimum of six months' time after approval of synopsis.

Sample Size: A sample size of 160 patients (80 exposed, 80 non-exposed) is calculated using 5% level of significance, 80% power of test. The frequency of UTI was taken as 30% in preeclampsia group and 12.1% in non-preeclampsia group.

Sampling technique: Non-probability consecutive sampling Inclusion Criteria

1. Patients attending OPD for routine antenatal checkup. 2. Patients with UTI as per operational definitions. 3. Patients with gestational age >20 weeks as per LMP 4. Age range of 18 to 35 years Exclusion Criteria

1. Patients with history of medical conditions like diabetes mellitus, chronic hypertension, chronic liver or kidney diseases, chronic pulmonary conditions.
2. Patients with history of urological surgical interventions in past 3 months.
3. Patients with history of renal transplants.
4. Patients on immunosuppression.
5. Patients with history of comorbid conditions like diabetes mellites, gestational diabetes mellitus, hypertension, chronic hepatic diseases, chronic liver diseases, chromic pulmonary diseases and ischemic heart diseases.
6. Patients with history of drugs intake during last one month which can cause proteinuria (NSAIDS, chemotherapeutic drugs, hydralazine, angiotensin receptor blockers).
7. Patients with a history of coagulation disorders.
8. Patients who are not willing for consent.

Data Collection Procedure:

After the study approval from the Ethical Review Committee, 160 women (80 exposed, 80 non-exposed) will be selected from the OPD of Obstetrics, PAF Hospital, Islamabad after fulfilling the required selection criteria. All the patients will be counselled regarding the research protocol and informed written consent will be obtained. All patients will undergo clinical evaluation and relevant investigations. Pregnant women will be instructed to collect their midstream urine sample in a sterile, wide-mouth container, approximately 10 ml, after washing their hands with water and cleaning their genital area using a swab soaked in normal saline. All samples will either be sent to the laboratory within 2 hours or stored in a refrigerator at 4°C and delivered to the laboratory within 18 hours of collection. The patients will be labelled as having UTI (exposed) and not having UTI (non-exposed) based on the operational definitions. The sampling process will continue until both groups have equal number of patients. All the patients will be followed until the parturition. The assessment will be done for the frequency of pre-eclampsia as per operational definitions. The assessment will be made by the consultant who will be kept blind of the exposed/unexposed groups. All patients will be managed as per hospital standard protocols. The results and respective data will be noted down on specially designed proforma attached as Annexure A.

DATA ANALYSIS The data will be analyzed by Statistical package for social sciences (SPSS) version 25 registered for Microsoft Windows. The quantitative variables like age, gestational age, BMI will be expressed as mean ± SD. The quantitative variables like parity, presence of UTI, preeclampsia will be expressed as frequency and percentages. The relative risk (RR) will be calculated for the development of preeclampsia in exposed and non-exposed groups. The data will be stratified for the effect modifiers like age, gestational age ang BMI. The post stratification RR will be recalculated. RR>1 and P value ≤ 0.05 will be considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending OPD for routine antenatal checkup
* Patients diagnosed with UTI as per operational definitions
* Gestational age greater than 20 weeks as per LMP
* Age between 18 to 35 years

Exclusion Criteria:

* History of medical conditions such as:
* Diabetes mellitus
* Chronic hypertension
* Chronic liver or kidney diseases
* Chronic pulmonary conditions
* History of urological surgical interventions in the past 3 months
* History of renal transplants
* Patients on immunosuppressive therapy
* History of comorbid conditions including:
* Diabetes mellitus
* Gestational diabetes mellitus
* Hypertension
* Chronic hepatic diseases
* Chronic liver diseases
* Chronic pulmonary diseases
* Ischemic heart diseases

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with gestational amenorrhea coming for routine antenatal checkup
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Preeclampsia | 37 weeks of pregnancy
  It will be defined as BP >140/90 mmHg on minimum two occasions after 20 weeks of pregnancy alongside presence of proteinuria (≥300 mg/day or at least 1+ dipstick testing or spot urine protein/creatinine ratio of ≥30 mg/mmol).

CONTACTS AND LOCATIONS:
Locations (1):
- PAF Hospital, Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson CY, Rocheleau CM, Howley MM, Chiu SK, Arnold KE, Ailes EC. Characteristics of Women with Urinary Tract Infection in Pregnancy. J Womens Health (Larchmt). 2021 Nov;30(11):1556-1564. doi: 10.1089/jwh.2020.8946. Epub 2021 Sep 1. PMID 34491115
- [Background] Haghdoost S, Pazandeh F, Khabazkhoob M, Bhroozi R. Assocoation Between Sexual and Genital Hygiene Habits with the Urinary Tact Infectin During Pregnancy: A Case-Control Study. International Journal of Women's Health and Reproduction Sciences. 2020;8(2):158-63.
- [Background] Radu VD, Vicoveanu P, Carauleanu A, Adam AM, Melinte-Popescu AS, Adam G, Onofrei P, Socolov D, Vasilache IA, Harabor A, Melinte-Popescu M, Scripcariu IS, Mihalceanu E, Stuparu-Cretu M, Harabor V. Pregnancy Outcomes in Patients with Urosepsis and Uncomplicated Urinary Tract Infections-A Retrospective Study. Medicina (Kaunas). 2023 Dec 7;59(12):2129. doi: 10.3390/medicina59122129. PMID 38138232
- [Background] Kaduma J, Seni J, Chuma C, Kirita R, Mujuni F, Mushi MF, van der Meer F, Mshana SE. Urinary Tract Infections and Preeclampsia among Pregnant Women Attending Two Hospitals in Mwanza City, Tanzania: A 1:2 Matched Case-Control Study. Biomed Res Int. 2019 Mar 27;2019:3937812. doi: 10.1155/2019/3937812. eCollection 2019. PMID 31032344
- [Background] Stitterich N, Shepherd J, Koroma MM, Theuring S. Risk factors for preeclampsia and eclampsia at a main referral maternity hospital in Freetown, Sierra Leone: a case-control study. BMC Pregnancy Childbirth. 2021 Jun 2;21(1):413. doi: 10.1186/s12884-021-03874-7. PMID 34078312
- [Background] Yaqub U, Khattak SN, Khattak MI, Akram U, Gardezi A, Mansoor K. Maternal Urinary Tract Infection and Risk of Preeclampsia: A Cross Sectional Comparative Study. J Soc Obstet Gynaecol Pak. 2022;12(1):1-6.
- [Background] Taghavi Zahedkalaei A, Kazemi M, Zolfaghari P, Rashidan M, Sohrabi MB. Association Between Urinary Tract Infection in the First Trimester and Risk of Preeclampsia: A Case-Control Study. Int J Womens Health. 2020 Jul 10;12:521-526. doi: 10.2147/IJWH.S256943. eCollection 2020. PMID 32765118
- [Background] Bajwa FA, Sultana N, Sadaqat A, Riaz A, Sikandar MZ. Factors contributing to preterm birth in patients presenting at tertiary care hospitals in Punjab. J Pak Med Assoc. 2024 Mar;74(3):504-508. doi: 10.47391/JPMA.9474. PMID 38591287
- [Background] Getaneh T, Negesse A, Dessie G, Desta M, Tigabu A. Prevalence of Urinary Tract Infection and Its Associated Factors among Pregnant Women in Ethiopia: A Systematic Review and Meta-Analysis. Biomed Res Int. 2021 Dec 1;2021:6551526. doi: 10.1155/2021/6551526. eCollection 2021. PMID 34901276
- [Background] Ghouri F, Hollywood A, Ryan K. Urinary tract infections and antibiotic use in pregnancy - qualitative analysis of online forum content. BMC Pregnancy Childbirth. 2019 Aug 13;19(1):289. doi: 10.1186/s12884-019-2451-z. PMID 31409404